CLINICAL TRIAL: NCT01771653
Title: Comparison of Two Triple Regimens for Treatment and Retreatment of Chronic Hepatitis C Infection
Status: Completed | Type: Observational
Sponsor: Southern Illinois University (Other)
Responsible Party: Sponsor
Other Study IDs: KOI-SIUSOM-12-002
Record Dates: First submitted 2013-01-16; First posted 2013-01-18 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Hepatitis C Infection
Keywords: Hepatitis C infection; Hepatitis C Virus; HCV
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Previously treated: Data from patients who were previously treated with Peg, interferon (IFN), alfa, and ribavirin
- Previously untreated: Records of patients who have never received anti-HCV treatment.

SUMMARY:
The purpose of this observational study is to compare two approved treatment regimen(s) containing boceprevir and telaprevir, as part of standard of care for the treatment of hepatitis C.

DETAILED DESCRIPTION:
The objective of the study is to compare the effect of adding 2 oral hepatitis C virus (HCV) protease inhibitors, telaprevir versus boceprevir, as part of current standard treatment regimen with (pegylated-interferon-alpha + ribavirin) for HCV Genotype-1 infection. Data will be obtained from medical records of consenting patients.

ELIGIBILITY:
Inclusion Criteria:

* Age - 18-64 years
* HCV genotype 1
* HCV RNA >100,000
* Liver biopsy within 5 years before enrollment
* Absolute neutrophil count of at least 1200 per cubic millimeter
* Platelet count of at least 90,000 per cubic millimeter
* Hemoglobin level of at least 12 g per deciliter
* Signed informed consent and Health Insurance Portability and Accountability Act (HIPAA) forms

Exclusion Criteria:

* HCV genotypes other than genotype 1
* Immunocompromised conditions including HIV, transplant or immunosuppressive drugs
* Decompensated liver disease or hepatocellular carcinoma
* Any other types of active cancer
* Active autoimmune disorders
* Major psychiatric disorders
* Active drug or alcohol use
* Pregnancy or lactation
* Patients with allergy to any of the drugs used in this study
* Drugs that may interact with boceprevir or telaprevir as listed in the package insert

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Population of adults aged 18-64 years, diagnosed with HCV genotype 1, with an HCV RNA >100,000. They should have had a liver biopsy within 5 years before enrollment. Lab work to determine eligibility includes an absolute neutrophil count of at least 1200 per cubic millimeter, a platelet count of at least 90,000 per cubic millimeter and a hemoglobin level of at least 12 g per deciliter
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2011-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Virologic Response | up to 96 weeks post treatment
  Sustained Virologic Response (SVR) rates will be compared between the two arms of treatment through measured HCV RNA levels after 24 weeks, 48 weeks and 96 weeks after completion of treatment.

SECONDARY OUTCOMES:
Adverse events | 24, 48, and 96 weeks post treatment
  Comparison of rates and severity of adverse events between the two study arms
Effect of baseline variables on treatment outcome | 24, 48, and 96 weeks post treatment
  Analyze the effects of baseline variables on treatment outcome between the two groups- age, race, social economic status.

CONTACTS AND LOCATIONS:
Overall Officials: Janak Koirala, MD, MPH, Principal Investigator — Southern Illinois University School of Medicine
Locations (1):
- Southern Illinois University School of Medicine, Springfield, Illinois, United States

REFERENCES:
- [Background] Lauer GM, Walker BD. Hepatitis C virus infection. N Engl J Med. 2001 Jul 5;345(1):41-52. doi: 10.1056/NEJM200107053450107. No abstract available. PMID 11439948
- [Background] Di Bisceglie AM, Lyra AC, Schwartz M, Reddy RK, Martin P, Gores G, Lok AS, Hussain KB, Gish R, Van Thiel DH, Younossi Z, Tong M, Hassanein T, Balart L, Fleckenstein J, Flamm S, Blei A, Befeler AS; Liver Cancer Network. Hepatitis C-related hepatocellular carcinoma in the United States: influence of ethnic status. Am J Gastroenterol. 2003 Sep;98(9):2060-3. doi: 10.1111/j.1572-0241.2003.t01-1-07641.x. PMID 14499788
- [Background] Witthoeft T, Hueppe D, John C, Goelz J, Heyne R, Moeller B, Teuber G, Wollschlaeger S, Baumgarten A, Simon KG, Moog G, Dikopoulos N, Mauss S. Efficacy and tolerability of peginterferon alfa-2a or alfa-2b plus ribavirin in the daily routine treatment of patients with chronic hepatitis C in Germany: the PRACTICE study. J Viral Hepat. 2010 Jul;17(7):459-68. doi: 10.1111/j.1365-2893.2009.01255.x. Epub 2010 Feb 11. PMID 20158603
- [Background] O'Brien TR, Everhart JE, Morgan TR, Lok AS, Chung RT, Shao Y, Shiffman ML, Dotrang M, Sninsky JJ, Bonkovsky HL, Pfeiffer RM; HALT-C Trial Group. An IL28B genotype-based clinical prediction model for treatment of chronic hepatitis C. PLoS One. 2011;6(7):e20904. doi: 10.1371/journal.pone.0020904. Epub 2011 Jul 8. PMID 21760886
- [Background] Poordad F, McCone J Jr, Bacon BR, Bruno S, Manns MP, Sulkowski MS, Jacobson IM, Reddy KR, Goodman ZD, Boparai N, DiNubile MJ, Sniukiene V, Brass CA, Albrecht JK, Bronowicki JP; SPRINT-2 Investigators. Boceprevir for untreated chronic HCV genotype 1 infection. N Engl J Med. 2011 Mar 31;364(13):1195-206. doi: 10.1056/NEJMoa1010494. PMID 21449783
- [Background] Koirala J, Gandotra SD, Rao S, Sangwan G, Mushtaq A, Htwe TH, Adamski A, Blessman D, Khardori NM. Granulocyte colony-stimulating factor dosing in pegylated interferon alpha-induced neutropenia and its impact on outcome of anti-HCV therapy. J Viral Hepat. 2007 Nov;14(11):782-7. doi: 10.1111/j.1365-2893.2007.00870.x. PMID 17927614
- [Background] Bacon BR, Gordon SC, Lawitz E, Marcellin P, Vierling JM, Zeuzem S, Poordad F, Goodman ZD, Sings HL, Boparai N, Burroughs M, Brass CA, Albrecht JK, Esteban R; HCV RESPOND-2 Investigators. Boceprevir for previously treated chronic HCV genotype 1 infection. N Engl J Med. 2011 Mar 31;364(13):1207-17. doi: 10.1056/NEJMoa1009482. PMID 21449784
- [Background] Jacobson IM, McHutchison JG, Dusheiko G, Di Bisceglie AM, Reddy KR, Bzowej NH, Marcellin P, Muir AJ, Ferenci P, Flisiak R, George J, Rizzetto M, Shouval D, Sola R, Terg RA, Yoshida EM, Adda N, Bengtsson L, Sankoh AJ, Kieffer TL, George S, Kauffman RS, Zeuzem S; ADVANCE Study Team. Telaprevir for previously untreated chronic hepatitis C virus infection. N Engl J Med. 2011 Jun 23;364(25):2405-16. doi: 10.1056/NEJMoa1012912. PMID 21696307
- [Background] Zeuzem S, Andreone P, Pol S, Lawitz E, Diago M, Roberts S, Focaccia R, Younossi Z, Foster GR, Horban A, Ferenci P, Nevens F, Mullhaupt B, Pockros P, Terg R, Shouval D, van Hoek B, Weiland O, Van Heeswijk R, De Meyer S, Luo D, Boogaerts G, Polo R, Picchio G, Beumont M; REALIZE Study Team. Telaprevir for retreatment of HCV infection. N Engl J Med. 2011 Jun 23;364(25):2417-28. doi: 10.1056/NEJMoa1013086. PMID 21696308
- [Background] McHutchison JG, Manns MP, Muir AJ, Terrault NA, Jacobson IM, Afdhal NH, Heathcote EJ, Zeuzem S, Reesink HW, Garg J, Bsharat M, George S, Kauffman RS, Adda N, Di Bisceglie AM; PROVE3 Study Team. Telaprevir for previously treated chronic HCV infection. N Engl J Med. 2010 Apr 8;362(14):1292-303. doi: 10.1056/NEJMoa0908014. PMID 20375406
- See also: telaprevir prescribing information — http://pi.vrtx.com/files/uspi_telaprevir.pdf